CLINICAL TRIAL: NCT00281021
Title: Phase II Trial of Second Line Erlotinib + Digoxin in Patients With Non-Small Cell Lung Cancer
Brief Title: Second Line Erlotinib (Tarceva) Plus Digoxin in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis revealed that only 1 patient had a partial response.
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Goetz Kloecker, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 629.05; BCC-LUN-05-001 (Other: James Graham Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: non-small cell lung cancer; Erlotinib; Digoxin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib and Digoxin (Experimental): Erlotinib plus Digoxin
  Interventions: Drug: Erlotinib plus Digoxin

INTERVENTIONS:
Drug: Erlotinib plus Digoxin — Each subject will receive erlotinib and digoxin daily until progression.
  Other Names: Tarceva; Digitalis

SUMMARY:
The purpose of this study is to determine the potential benefit of adding Digoxin to erlotinib (Tarceva) treatment for patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) accounts for 80% of all lung cancer cases. The majority of NSCLC patients have advanced disease at the time of diagnosis, which usually requires treatment beyond standard first-line chemotherapy. Until recently, patients were limited in the number of options available for second-line treatment of NSCLC. In 2004, erlotinib was approved by the FDA for second and third-line treatment of NSCLC. Erlotinib is a cancer chemotherapy medication that slows the growth and spread of cancer cells in the body.

Recent research suggests that a medication called Digoxin can sensitize cancer cells to respond better to chemotherapy. Digoxin is normally used to treat certain heart conditions by helping the heart beat more strongly and regularly and is not approved by the FDA for the treatment of NSCLC. Investigators hope that subject response rates to standard erlotinib therapy will be significantly improved by the addition of Digoxin.

The purpose of this study is to determine the tumor response rate and overall survival of patients with non-small cell lung cancer treated with a daily regimen of erlotinib (Tarceva) plus Digoxin.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of non-small cell lung cancer
* measurable or evaluable disease
* primary tumor must be documented by histopathic analysis
* disease recurrences occurring greater than five years after original diagnosis must be biopsy proven
* treatment with only one prior chemotherapy regimen for advanced disease (one additional prior regimen was allowed for neoadjuvant, adjuvant, or neoadjuvant plus adjuvant therapy)
* serum creatinine < 2mg/dl, or a calculated creatinine clearance > 40cc/min using the following formula: (140-age) x WT(kg) x 0.85 (if female 0.72) x creatinine (mg/dl). Tests must be done within 28 days prior to registration
* must have a CT scan (chest & abdomen) within 4 weeks prior to registration
* Zubrod performance status of 0-3

Exclusion Criteria:

* women who are pregnant or nursing
* no other prior malignancy is allowed except for: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* history of ventricular fibrillation, sinus node or AV nodal disease, Wolff Parkinson White Syndrome, evidence of congestive heart failure, chest pain with exertion, hemodynamically significant or life threatening cardiac arrhythmia, or evidence of prior myocardial infarction on EKG. EKG must have been done within 28 days prior to registration. A normal cardiac stress test within 182 days prior to registration is required for all patients over 50 years old or those with abnormal EKG or any history of cardiac disease.
* hypersensitivity to erlotinib and/or Digoxin
* abnormal levels of K, Mg, and/or Ca, or conditions which cause such abnormalities (e.g. malnutrition, severe diarrhea, prolonged vomiting, dialysis, GI suction, untreated hypothyroidism, and use of diuretics, amphotericin B, steroids, or antacids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, MSPH, Principal Investigator — James Graham Brown Cancer Center/ University of Louisville

REFERENCES:
- See also: James Graham Brown Cancer Center — http://www.browncancercenter.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient accrual lasted from March 2006 until August 2008 and was stopped early at the time of interim analysis. 24 who completed at least 6 weeks of therapy are presented here.
Groups:
- Erlotinib and Digoxin: Erlotinib plus Digoxin
  Erlotinib plus Digoxin : Each subject will receive erlotinib and digoxin daily until progression.
Period: Overall Study
Arm/Group | Erlotinib and Digoxin
Started | 26
Completed | 24
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib and Digoxin
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 61 [34 to 78]
Age, Customized [Number; unit: participants]
  <=18 years | 0
  >18 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Response, Evaluated by Computed Tomography (CT) Scans of Chest & Abdomen.
Time Frame: Measured every 6 weeks after baseline until disease progression, an average of 3 months
Measure: Number; unit: participants
Arm/Group | Erlotinib and Digoxin
Number analyzed (Participants) | 24
participants
  Partial Response | 1
  Stable Disease | 9
  Progressive Disease | 14

ADVERSE EVENTS:
Arm/Group | Erlotinib and Digoxin
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 20/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Digoxin (N=24)
Diarrhea (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 5
Rash (General disorders) | 10
Nausea (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes